CLINICAL TRIAL: NCT04990479
Title: An Open-Label, Multicenter, Non-Randomized, Dose-Confirmation and Cohort-Expansion Phase 1b Study to Evaluate the Safety, Tolerability, and Anti-Tumor Activity of Nous-PEV, with Pembrolizumab, in Patients with Unresectable Stage III / IV Cutaneous Melanoma and with Stage IV NSCLC (PDL1≥ 50%)
Brief Title: Nous-PEV: a Novel Immunotherapy for Lung Cancer and Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Nouscom SRL (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOUS-PEV-01; 2019-004759-35 (EudraCT Number)
Record Dates: First submitted 2021-07-15; First posted 2021-08-04 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Melanoma (Skin); Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Treatment Cohorts of the study.
  Part 1:
  • Cohort 1a: 3 patients (expandable to 9) with unresectable stage III / IV Cutaneous Melanoma.
  Part 2
  * Cohort 2a: 13 patients with unresectable stage III / IV Cutaneous Melanoma.
  * Cohort 2b:12 patients with stage IV NSCLC (PDL1≥ 50%). In all cohorts, the treatment consists of four Nous-PEV vaccine administrations in combination with pembrolizumab as SoC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1a (Experimental): Cohort 1a: 3 patients (expandable to 9) with unresectable stage III / IV Cutaneous Melanoma.
  Interventions: Biological: GAd-PEV; Biological: MVA-PEV
- Cohort 2a (Experimental): Cohort 2a:13 patients with unresectable stage III / IV Cutaneous Melanoma.
  Interventions: Biological: GAd-PEV; Biological: MVA-PEV
- Cohort 2b (Experimental): Cohort 2b: 12 patients with stage IV NSCLC (PDL1≥ 50%).
  Interventions: Biological: GAd-PEV; Biological: MVA-PEV

INTERVENTIONS:
Biological: GAd-PEV — Priming phase including 1 GAd-PEV administration with Standard of Care pembrolizumab (cycle 4).
Biological: MVA-PEV — Boosting phase including 3 boosting administrations of MVA-PEV with Standard of Care pembrolizumab (cycles 5, 6 and 7).

SUMMARY:
From Protocol v3.0 dated 16Jun2022. This is an international, multicenter, open-label, multiple cohort, First in Human, phase 1b clinical study, designed to evaluate safety, tolerability, and immunogenicity, and to detect any preliminary evidence of anti-tumor activity of a personalized vaccine (PEV) based on GAd-PEV priming and MVA-PEV boosting, combined with SoC first-line immunotherapy using an anti-PD-1 checkpoint inhibitor in patients with unresectable stage III/IV cutaneous melanoma or with stage IV NSCLC (PDL1 ≥ 50%). The PEV vaccines will be prepared on an individual basis, following a tumor biopsy performed at the time of screening and subsequent NGS analysis, to identify patient-specific tumor mutations. Both neoantigen-encoding genetic vaccines are administered intramuscularly using 1 prime with GAd-PEV and 3 boosts with MVA-PEV in combination with the licensed programmed death receptor-1 (PD-1)-blocking antibody pembrolizumab in adult patients in patients with unresectable stage III/IV cutaneous melanoma (Cohort a) or with stage IV NSCLC (PDL1 ≥ 50%) (Cohort b).

DETAILED DESCRIPTION:
Overall Study Design:

• This is an open-label, non-randomized, dose-confirmation and cohort expansion phase 1b first-in-human study, in which 28 patients, expandable up to 34 evaluable patients in case of DLT.

Study IMPs:

Nous-PEV vaccine is composed of 2 sets of IMPs:

* GAd-PEV
* MVA-PEV

Treatment phases:

A) Induction phase with pembrolizumab (cycles 1, 2 and 3). B) Priming phase including 1 GAd-PEV administration with pembrolizumab (cycle 4).

C) Boosting phase including 3 boosting administrations of MVA-PEV with pembrolizumab (cycles 5, 6 and 7).

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria for Patients in Cohorts 1a and 2a:

1. Age ≥ 18 years.
2. Patients with histologically or cytologically confirmed unresectable stage III or stage IV Cutaneous Melanoma, as per AJCC staging system (8th edition). First-line treatment-naive patients.
3. Participation in this trial will be dependent upon supplying tumor tissue from newly obtained specimen. Newly obtained biopsies of a tumor lesion, not previously irradiated, must be provided in the form of excisional biopsies, resected tissue or core needle biopsies.
4. Presence of at least 1 measurable lesion by computed tomography or magnetic resonance imaging per RECIST v1.1 by the local site Investigator / radiologist assessment
5. Presence of at least one lesion amenable to repeated biopsy, ideally not the one being used for measuring.
6. Willingness to undergo a minimum of two fresh lesion biopsies (pre-treatment and on-treatment).
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
8. Life expectancy of at least 12 months.
9. Adequate renal, hepatic, and hematologic functions
10. A female patient is eligible to participate if she is not pregnant and not breastfeeding
11. A male patient must agree to use an adequate contraception

Main Inclusion Criteria for Patients in Cohort 2b:

1. Age ≥ 18 years.
2. Histologically or cytologically confirmed stage IV squamous or non-squamous NSCLC without EGFR or ALK/ROS1 /RET genomic alteration.
3. Tumor expression with PD-L1 ≥50% tumor proportion score (TPS).
4. First-line treatment-naïve patients.
5. Participation in this trial will be dependent upon supplying tumor tissue from a newly obtained specimen. Newly obtained biopsies of a tumor lesion, not previously irradiated, must be provided in the form of excisional biopsies, resected tissue or core needle biopsies.
6. Presence of at least 1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST v1.1 as determined by the local site Investigator / radiologist assessment.
7. Presence of at least one tumor lesion amenable to repeated biopsy, if possible, ideally not the one being used for measuring.
8. Willingness to undergo a minimum of two fresh tumor biopsies (pre-treatment and on-treatment).
9. ECOG performance status 0 to 1.
10. Life expectancy of at least 6 months.
11. Adequate renal, hepatic, and hematologic functions
12. A female patient is eligible to participate if she is not pregnant and not breastfeeding
13. A male patient must agree to use a contraceptive during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.

Main Exclusion Criteria for patients in all Cohorts:

1. Currently receiving treatment with another investigational medicinal product.
2. Prior therapy with immune checkpoint inhibitors. Patients must not have received any investigational immunotherapy either.
3. Prior radiotherapy within 2 weeks of enrolment, or within 4 weeks of enrolment in the case of radiation to central nervous system (CNS), which requires ≥ 4-week washout.
4. Prior allogenic tissue or solid organ transplant.
5. Active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring treatment with systemic steroids and/or whose pulse oximetry is less than 92% "on room air".
6. Limiting cardiac criteria: prolonged QT interval or QT prolongation risk factors, clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g. complete LBBB, third degree heart block, risk of arrythmic events, ejection fraction under lower limit of normal.
7. Major (according to the Investigator's judgment) surgery within 12 weeks before enrolment.
8. Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry.
9. Immunosuppression including the continued use of systemic (at prednisone dose equivalent of > 10 mg) or topical steroids at or near the planned i.m. injection site or the use of immunosuppressive agents for any concurrent condition in the 4 weeks prior to first study treatment administration. Inhaled and eye drop-containing corticosteroids are permitted.
10. Previous vaccination (either therapeutic and/or prophylactic) against cancer.
11. History of autoimmune disease in the last 5 years, including any active autoimmune disease except vitiligo or childhood asthma.
12. Chronic or concurrent active infectious disease requiring systemic antibodies, antifungal, or antiviral treatment.
13. Known Medical History of human immunodeficiency virus (HIV) infection or known Medical History of acquired immunodeficiency syndrome (AIDS). HIV testing is not required unless mandated by the local health authority.
14. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection that requires treatment, or at risk for HBV reactivation
15. Known CNS metastasis and/or carcinomatous meningitis.
16. Known cerebral edema.
17. Live vaccine received within 30 days before treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: incidence of treatment- emerging adverse events. AEs characterized by type, severity (graded by CTCAE v.5.0), Timing, seriousness and relationship to study treatments. | Up to 110 weeks
  * Frequency, duration, and severity of adverse events (AEs) and serious adverse events (SAEs) using CTCAE v5.0 criteria.
  * Changes in vital signs and clinical evaluations.
  * Changes in clinical laboratory blood samples.
  * Dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
RP2D confirmation 2. Clinical efficacy: | Up to 110 weeks
  RP2D confirmation based on safety and tolerability
Clinical efficacy | Up to 110 weeks
  Clinical efficacy based on Overall response rate (ORR); Best overall response (BOR); Duration of response (DoR); Progression-free survival (PFS); Overall survival (OS), all as defined in tumor imaging, RECIST 1.1

OTHER OUTCOMES:
Exploratory outcome: immunogenicity | Up to 110 weeks
  PBMC-derived T-cell responses against vaccine FSPs, as measured by IFN-gamma ELISpot

CONTACTS AND LOCATIONS:
Overall Officials: Sven Gogov, MD, Study Director — Nouscom SRL
Locations (7):
- Belgium (2):
  - Grand Hopital de Charleroi, Grand Rue 3, 6000 Charleroi, Charleroi
  - UZ Leuven Hospital, Campus Gasthuisberg, Herestraat 49, 3000 Leuven, Leuven
- Spain (4):
  - Institut Catalá d'Oncologia ICO L'Hospitalet. Av Gran Via de L'Hospitalet 199-203. 08908 L'Hospitalet de Llobregat, Barcelona, Spain, Barcelona
  - START Madrid - Centro Integral Oncológico Clara Campal, HM CIOCC Hospital Universitario HM Sanchinarro, 28050 Madrid. Spain, Madrid
  - START Madrid-FJD, Hospital Fundación Jiménez Diaz Avda. Reyes Católicos 2. 28040, Madrid, Spain, Madrid
  - Instituto de Investigación Sanitaria INCLIVA - Hospital Clínico Universitario de Valencia. Av. Blasco Ibáñez, 17 CP 46010 Valencia, Spain, Valencia
- Cancer Research UK Edinburgh Centre. Western General Hospital, Edinburgh, EH4 2SP, UK, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leoni G, D'Alise AM, Tucci FG, Micarelli E, Garzia I, De Lucia M, Langone F, Nocchi L, Cotugno G, Bartolomeo R, Romano G, Allocca S, Troise F, Nicosia A, Lahm A, Scarselli E. VENUS, a Novel Selection Approach to Improve the Accuracy of Neoantigens' Prediction. Vaccines (Basel). 2021 Aug 9;9(8):880. doi: 10.3390/vaccines9080880. PMID 34452005
- [Derived] D'Alise AM, Leoni G, Cotugno G, Siani L, Vitale R, Ruzza V, Garzia I, Antonucci L, Micarelli E, Venafra V, Gogov S, Capone A, Runswick S, Martin-Liberal J, Calvo E, Moreno V, Symeonides SN, Scarselli E, Bechter O. Phase I Trial of Viral Vector-Based Personalized Vaccination Elicits Robust Neoantigen-Specific Antitumor T-Cell Responses. Clin Cancer Res. 2024 Jun 3;30(11):2412-2423. doi: 10.1158/1078-0432.CCR-23-3940. PMID 38506710
- See also: VENUS is a proprietary algorithm designed to enhance the predictive accuracy of personalized neoantigen selection, used in the NOUS-PEV-01 trial. — https://pubmed.ncbi.nlm.nih.gov/34452005/